CLINICAL TRIAL: NCT03802253
Title: Study to Evaluate the Effects of Time-Restricted Feeding Regimen in Overweight/Obese Subjects With Impaired Glucose Regulation
Brief Title: Time Restricted Feeding on Impaired Glucose Regulation(TRIG Trial)
Acronym: TRIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KYH2019-001
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Time-Restricted Feeding; Impaired Glucose Regulation; Overweight/Obese
MeSH Terms: conditions — Intermittent Fasting; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRF (Experimental): Participants in this group will focus on time restricted feeding (TRF) in addition to daily calorie restriction.
  Interventions: Behavioral: Time Restricted Feeding(TRF)
- RCD (Active Comparator): Participants in this group will focus on standard care with daily reduced calorie diet (RCD)
  Interventions: Behavioral: Reduced Calorie Diet (RCD)

INTERVENTIONS:
Behavioral: Time Restricted Feeding(TRF) — Participants will receive a diet of 1200-1500kcal/d and be instructed to eat only during a window of 8 hours (Finishing the last meal before 4pm) in the first 6 months. 6 months later, Participants will receive a diet of 1200-1500kcal/d without a restriction of feeding time.
  Arms: TRF
Behavioral: Reduced Calorie Diet (RCD) — Participants will receive a diet of 1200-1500kcal/d and keep their usual eating pattern.
  Arms: RCD

SUMMARY:
We evaluated the effects of Time-Restricted Feeding (TRF) regimen on Impaired Glucose Regulation (IGR) in comparison with overweight/obese patients receiving standard of care over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 year
2. Diagnosis of impaired glucose regulation (i.e. FG between 5.7-6.9mmol/L) +/- impaired glucose tolerance (i.e. 2-hour postprandial PG between 7.8-11.1mmol/L) confirmed by latest OGTT results within 3 months prior to recruitment
3. Body mass index (BMI)of 23.0 to 45.0 kg/m2;

Exclusion Criteria:

1. Confirmed diagnosis of DM or on hypoglycaemic treatment
2. Women who are pregnant or breast-feeding at recruitment
3. Patients taking glucocorticoid at recruitment
4. Active and uncontrolled thyroid diseases (including subjects on thyroid replacement therapy or anti-thyroid drugs) or active endocrine diseases such as Cushing's syndrome or Acromegaly at recruitment
5. Serious liver dysfunction or chronic kidney disease (AST or ALT > 3 times the upper limit of normal, or eGFR<30 ml/min/1.73 m2);
6. History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
7. Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
8. Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight) ;
9. Patients who cannot be followed for 24 months (due to a health situation or migration);
10. Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c level (%) | 3 months, 6 months and 12 months
Change in serum fasting insulin levels (pmol/L) | 3 months, 6 months and 12 months
Incidence of regression to normoglycaemia among the studied population | 12 months

SECONDARY OUTCOMES:
Changes in body weight (Kilograms) | 3 months, 6 months and 12 months
Changes in waist circumference (cm) | 3 months, 6 months and 12 months
Change in body mass index (kg/m2) | 3 months, 6 months and 12 months
Changes in systolic pressure (mmHg) | 3 months, 6 months and 12 months
Changes in diastolic pressure (mmHg） | 3 months, 6 months and 12 months
Changes in fasting blood glucose (mmol/L) | 3 months, 6 months and 12 months
Change in β cell function | 3 months, 6 months and 12 months
  β cell function will be assessed by HOMA-β
Change in insulin sensitivity | 3 months, 6 months and 12 months
  Insulin sensitivity will be assessed by HOMA-IR
Changes in serum total cholesterol levels (mmol/L) | 3 months, 6 months and 12 months
Changes in serum low density lipoprotein cholesterol levels (mmol/L) | 3 months, 6 months and 12 months
Changes in serum triglyceride levels (mmol/L) | 3 months, 6 months and 12 months
Changes in serum high density lipoprotein cholesterol levels (mmol/L) | 3 months, 6 months and 12 months
Changes in serum alanine aminotransferase levels levels (mmol/L) | 3 months, 6 months and 12 months
Changes in serum aspartate aminotransferase levels (mmol/L) | 3 months, 6 months and 12 months
Changes in serum gamma glutamyltranspeptidase levels (mmol/L) | 3 months, 6 months and 12 months
Changes in controlled attenuation parameter(dB/m) | 3 months, 6 months and 12 months
  Controlled attenuation parameter will be assessed by transient elastography (FibroScan(®) ）
Changes in Changes in liver fibrosis | 3 months, 6 months and 12 months
  Liver fibrosis will be assessed by transient elastography (FibroScan(®) ）
Changes in Epworth sleepiness scores（ESS) | 3 months, 6 months and 12 months
  The range of epworth sleepiness scores（ESS) is from 0 to 24 and higher scores mean worse outcome.
Changes in depressive symptoms | 3 months, 6 months and 12 months
  Depressive symptoms will be assessed by Patient Health Questionnaire-9 (PHQ-9) algorithm scoring method. The range of PHQ-9 is from 0 to 27 and higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Xiamen university, Xiamen, Fujian, China